CLINICAL TRIAL: NCT03156075
Title: Sponsor Investigator, Assistant Professor at Public Health and Community Medicine Department, Faculty of Medicine, Assiut University
Brief Title: Postoperative Intervention Program Effectiveness in Hip Fracture Patients: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalia Mahran (Other)
Responsible Party: Sponsor-Investigator, Dalia Mahran, Assistant professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17300078
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Hip Fractures
Keywords: hip fracture, intervention, mortality, mobility
MeSH Terms: conditions — Hip Fractures | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group will receive the nutrition and exercise program intervention. Nutrition education will be about increasing the intake calcium and vitamin D rich foods and exposure to sun will provided for the intervention group.
  Education of the patients about exercises that increases the strength of lower limb and hip muscles to increase the mobility of the patients earlier and decrease the mortality in turn.
  and the first one will start before discharge. The patients will receive a leaflet to describe the instructions.
  Interventions: Behavioral: Nutrition and exercise program
- Control group (No Intervention): This group will be selected from the previous three months, they didn't receive any intervention and received the usual care postoperative.

INTERVENTIONS:
Behavioral: Nutrition and exercise program — Nutrition education will be about increasing the intake calcium and vitamin D rich foods and exposure to sun will provided for the intervention group.
  Education of the patients about exercises that increases the strength of lower limb and hip muscles to increase the mobility of the patients earlier and decrease the mortality in turn.
  Arms: Intervention group

SUMMARY:
The aim of the study is to investigate whether a simple intervention improves the physical functioning and reduce mortality after surgery for elderly hip fracture patients in a period of one year follow up. We hypothesized that the postoperative intervention program decreases the mortality in one year and improves mobility.

This study is a randomized controlled trial designed as a prospective intervention and a historical control group from the previous three months admitted operated hip fracture patients from another study and with bone mineral density and measurement of weight and height done. The study will include patients of both sexes, 50 years and older, after their approval to participate and applying exclusion criteria. A baseline assessment will be done for the included hip fracture patients, who will be admitted to Trauma Unit of Assiut University Hospitals and will be surgically treated for a period of 1 year. The exclusion criteria include patients with major accidents, polytrauma, pathological fractures and bilateral hip fractures. Also patients with thyroid malfunctions, renal diseases, cardiac diseases, long term immobilization, liver diseases and musculoskeletal disorders. Two well-trained nurses will carry out the personal interviews in the Trauma Unit ward with each patient and/or patients 'relatives using a structured questionnaire. Data collection will be done after providing informed consent.

Bone mineral density, weight and height for every patient will be done. The follow up phone calls will be done for every patient at 3 months, 6 months and one year postoperative.

Intervention group:

Patients in the intervention Group will be provided with postoperative health education intervention program, which includes nutrition education for improving general and bone health and physical exercise training for the patient and his relative before discharge.

This group will receive the usual care prior to the start of intervention and participating in the study.

The phone calls will include questions about: if the patient is alive or not. If not, subsequent detailed questions about causes and timing of death will be filled in.

If the patient is alive, subsequent questions about nutrition, commodities and physical activity will be filled in. Assessment of physical activity will be done by the Western Ontario And McMaster Universities Osteoarthritis Index (WOMAC).

DETAILED DESCRIPTION:
The aim of the study is to investigate whether a simple intervention improves the physical functioning and reduce mortality after surgery for elderly hip fracture patients in a period of one year follow up. We hypothesized that the postoperative intervention program decreases the mortality in one year and improves mobility.

This study is a randomized controlled trial designed as a prospective intervention and a historical control group from the previous three months admitted operated hip fracture patients from another study and with bone mineral density and measurement of weight and height done.

The study will include patients of both sexes, 50 years and older, after their approval to participate and applying exclusion criteria. A baseline assessment will be done for the included hip fracture patients, who will be admitted to Trauma Unit of Assiut University Hospitals and will be surgically treated for a period of 1 year. We aim to minimize other factors that affect the intervention program compliance and could increase the mortality. The exclusion criteria include patients with major accidents, polytrauma, pathological fractures and bilateral hip fractures. Also patients with thyroid malfunctions, renal diseases, cardiac diseases, long term immobilization, liver diseases and musculoskeletal disorders.

Two well-trained nurses will carry out the personal interviews in the Trauma Unit ward with each patient and/or patients 'relatives using a structured questionnaire. Data collection will be done after providing informed consent. The questionnaire for baseline data includes sociodemographic characteristics such as name, sex, and age, associated comorbidities and some nutrition habits. The nutrition habits in pre and post intervention will be evaluated by the dietary history qualitative subjective method using closed ended questions [1].

Bone mineral density (BMD) evaluation and anthropometric measurements:

BMD measurements will be assessed as soon as possible postoperative for all participants by dual-energy x-ray absorptiometry (DEXA) scan of the femoral neck, using GE Lunar, GE Healthcare, USA.

From the measured BMD, sex-specific T scores will be calculated. All DEXA measurements will be carried out by one machine and the interpretations by the same radiologist. The criteria recommended by the International Osteoporosis Foundation and the World Health Organization were used to assess BMD and to determine the prevalence of osteoporosis. BMD will be assessed according to T score and classified to three groups as normal (T score ≥ -1 SD), osteopenic (T score from -1 to -2.5 SD), or osteoporotic (T score ≤ -2.5SD) [2]. Height while lying down without shoes and weight will be measured while the patients were dressed in light clothes. Body mass index (BMI) was calculated from the height and weight will be recorded while performing the DEXA scan. The BMI will be calculated based on the formula: weight (kg)/[height (m)]2. The standard categorization of BMI by Center for Disease Control and Prevention (CDC) indicates less than 18.5 as underweight, 18.5-24.9 as normal, 25.0-29.9 as overweight, and 30.0 and above as obese [3].

The data collectors will include patients from the prior three months that their DEXA and anthropometric measurements in addition to their telephone numbers were available, while the equal number of patients will be prospectively included in the intervention group during the period of the study.

An independent investigator, who will not involved with recruitment or data collection, a trained another team on the intervention program to conduct it for every selected patient.

The follow up phone calls will be done for every patient at 3 months, 6 months and one year postoperative. All calls will be done by one assessor; who will not be blinded to group allocation as the patients mentioned the intervention program during phone calls.

Intervention group:

Patients in the intervention Group (IG) will be provided with postoperative health education intervention program, which includes nutrition education for improving general and bone health and physical exercise training for the patient and his relative before discharge.

The Intervention Protocol:

Each patient and a family member will receive a 10-minute explanation about postoperative nutrition and physical exercise during their postoperative hospital stay. In addition, the patients will receive an explanatory leaflet of the health education messages to assure their continuity to follow the instructions after hospital discharge. Nutrition instructions includes instructions about habits and foods that augment calcium and vitamin D requirements and general health. All foods are public and inexpensive. For example increase the intake of milk products and eggs. Increase the duration of exposure to sun light will be advised. They will receive education messages about factors decreasing the calcium absorption as drinks with excess caffeine and carbonated soft.

Control group:

This group will receive the usual care prior to the start of intervention and participating in the study. Usual care is what the patient receives as part of the hospital standard care. Prescription of calcium and vitamin D will be done for all patients. No specific personal communication regarding nutrition or physical activity will be provided.

Follow up phone calls after intervention:

The phone calls with both groups will be done at 3 months, 6 months and one year postoperative by one assessor, A follow up questionnaire will be filled in by the assessor from the patient or his relative, who is responsible for the patient's care. The questionnaire consists of three sections, the first one is asking about the patient if she/he is alive or not. If she/he died, reason for death and duration from the operation till death will be inquired. The second section will be about the preoperative conditions as duration between the fracture and the index surgery and postoperative hospital stay. Also questions about the postoperative complications and health problems (pulmonary, cardiac, cerebrovascular stoke, urinary tract infections, depression and others). The third section is about applying the nutrition guides as stop smoking and drinking milk, eating cheese, yogurt and eggs. Regular intake of calcium and vitamin D supplements will be asked about. Maintenance and regularity of physical activity as in the provided instructions of the intervention postoperative care program.

Assessment of physical activity will be done by the Western Ontario And McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC has been validated for telephone assessment [4]. The WOMAC is available in over 65 alternate language forms, including Arabic [5], to assess pain, stiffness, and physical function in patients with hip and / or knee osteoarthritis (OA). The WOMAC consists of 24 items divided into 3 sub scales: 1- Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing. 2- Stiffness (2 items): morning stiffness after waking up and later in the day. 3- Physical Function includes 17 items. A total WOMAC score is created by summing the items for all three sub scales. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. Each item score ranged from 0-4 with total score of 96 (100%). Time to score was 10-15 minutes.

Statistical analysis will be carried out using the Statistical Package for the Social Sciences version 22 (SPSS Inc., Chicago, US).

ELIGIBILITY:
Inclusion Criteria:

All patients postoperative hip fracture from 50 years and above from both sexes and admitted to Trauma Unit at Assiut University Hospitals

Exclusion Criteria:

* patients with major accidents, polytrauma, pathological fractures and bilateral hip fractures. Also patients with thyroid malfunctions, renal diseases, cardiac diseases, long term immobilization, liver diseases and musculoskeletal disorders.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mortality | immediately postoperative to one year after operation
  Postoperative hip fracture mortality of the patients

SECONDARY OUTCOMES:
Mobility | from three months to one year postoperative
  Mobility of the patient to start independent painless improving movements to return to normal life

IPD SHARING:
Plan to Share IPD: No